CLINICAL TRIAL: NCT04442295
Title: An Open-Label Study to Investigate the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of Antisense Oligonucleotide STK-001 in Children and Adolescents With Dravet Syndrome
Brief Title: An Open-Label Study to Investigate the Safety of Single and Multiple Ascending Doses in Children and Adolescents With Dravet Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stoke Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STK-001-DS-101
Record Dates: First submitted 2020-06-08; First posted 2020-06-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Dravet Syndrome
Keywords: Pediatric epilepsy; Epileptic Encephalopathies; Refractory Myoclonic Epilepsy; Severe Myoclonic Epilepsy in Infancy
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Doses (Experimental): Enrollment of patients in two age groups. A Sentinel group of 2 patients aged 13 to 18 years of age, inclusive, and an expanded group of 2 patients 2 to 12 years of age to receive single doses. There will be an option to dose up to 6 additional patients at each dose level and an option to expand the maximum tolerated dose level with 5 additional patients.
  Interventions: Drug: STK-001 - Single Ascending Doses
- Multiple Ascending Doses (Experimental): Enrollment of patients in two age groups. A Sentinel group of 2 patients aged 13 to 18 years of age, inclusive, and an expanded group of 2 patients 2 to 12 years of age to receive multiple doses. There will be an option to dose up to 6 additional patients at each dose level and an option to expand the maximum tolerated dose level with 10 additional patients.
  Interventions: Drug: STK-001 - Multiple Ascending Doses

INTERVENTIONS:
Drug: STK-001 - Single Ascending Doses — Experimental : Single Ascending Doses - STK-001 drug product is an antisense oligonucleotide administered as an intrathecal injection. Four dose levels will be evaluated ( 10mg, 20mg,30mg, 45mg and 70mg ).
  Arms: Single Ascending Doses
Drug: STK-001 - Multiple Ascending Doses — Experimental : Multiple Ascending Doses - STK-001 drug product is an antisense oligonucleotide administered as an intrathecal injection. Three dose levels will be evaluated ( 20mg,30mg and 45mg ).
  Arms: Multiple Ascending Doses

SUMMARY:
Stoke Therapeutics is evaluating the safety and tolerability of single and multiple ascending doses of STK-001 in patients with Dravet syndrome. Change in seizure frequency, overall clinical status, and quality of life will be measured as secondary endpoints in this open-label study.

DETAILED DESCRIPTION:
STK-001 is an investigational new medicine for the treatment of Dravet syndrome. STK-001 is an antisense oligonucleotide (ASO) that is intended to increase the level of productive SCN1A messenger RNA (mRNA) and consequently increase the expression of the sodium channel Nav1.1 protein. This RNA-based approach is not gene therapy, but rather RNA modulation, as it does not manipulate nor insert genetic deoxyribonucleic acid (DNA).

STK-001 is designed to upregulate Nav1.1 protein expression from the nonmutant (wild-type) copy of the SCN1A gene to restore physiological Nav1.1 levels. Nav1.1 levels are reduced in people with Dravet syndrome. Stoke has generated preclinical data demonstrating proof-of-mechanism for STK-001.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Dravet Syndrome (DS) with onset of recurrent focal motor or hemiconvulsive or generalized tonic-clonic seizures prior to 12 months of age, which are often prolonged and triggered by hyperthermia.

  * No history of causal MRI lesion
  * No other known etiology
  * Normal development at seizure onset.
* Documented pathogenic, likely pathogenic variant, or variant of uncertain significance in the SCN1A gene associated with DS.
* Use of at least 2 prior treatments for epilepsy that either had lack of adequate seizure control (requiring an additional AED) or had to be discontinued due to an AE(s).
* Currently taking at least one AED at a dose which has been stable for at least 4 weeks prior to Screening.
* Stable epilepsy medications or interventions for epilepsy (including ketogenic diet or vagal nerve stimulator) for at least 4 weeks prior to Screening.

Exclusion Criteria:

* Known pathogenic mutation in another gene that causes epilepsy
* Currently treated with an AED acting primarily as a sodium channel blocker, as maintenance treatment, including: phenytoin, carbamazepine, oxcarbazepine, lamotrigine, lacosamide, or rufinamide.
* Clinically significant unstable medical conditions other than epilepsy.
* Clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to Screening or prior to dosing on Day 1, other than epilepsy.
* History of brain or spinal cord disease (other than epilepsy or DS), or history of bacterial meningitis or brain malformation
* Spinal deformity or other condition that may alter the free flow of cerebrospinal fluid (CSF) or has an implanted CSF drainage shunt.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, may influence the results of the study, or may affect the patient's ability to participate in the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of single and multiple doses of STK-001 with respect to: | Screening (Day -28) until 6 months after single and multiple drug dosing
  1. Incidence of adverse events
  2. incidence of abnormal vital signs
  3. Abnormal physical examination findings
  4. Abnormal 12-lead electrocardiogram (ECG)
  5. Abnormal laboratory parameters
Pharmacokinetic (PK) Parameters | Day 1 (Dosing) until 6 months after single and multiple drug dosing
  Analysis of plasma concentrations of STK-001
Exposure of STK-001 in Cerebrospinal Fluid (CSF) | Day 1 (Dosing) until 6 months after single and multiple drug dosing
  Measurement of STK-001 concentrations

SECONDARY OUTCOMES:
Measurement of seizure frequency | Screening (Day -28) until 6 months after single and multiple drug dosing
  Measured by paper diary
Change in Caregiver Global Impression of Change Scale | Baseline (Day -1) until 6 months after single and multiple drug dosing
  Change from baseline in overall clinical status as measured by the Clinical Global Impression of Change (CGIC).
  Values of scales:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Change in Clinician-assessed Global Impression of Change Scale | Baseline (Day -1) until 6 months after single and multiple drug dosing
  Change from baseline in overall clinical status as measured by the Caregiver Global Impression of Change (CaGIC)
  Values of scales:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Measurement of Quality of Life | Baseline (Day -1) until 6 months after single and multiple drug dosing
  Change in quality of life as measured by the EuroQoL-five dimensions, youth version (EQ-5D-Y) instrument. The scale is scored from 0-100. The reference to a high score indicates a better outcome of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Dandurand, MD, Study Director — Medical Director
Locations (18):
- United States (18):
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics; Pediatric Specialty Clinic, Iowa City, Iowa
  - Massachusetts General Hospital - Pediatric Epilepsy Program, Boston, Massachusetts
  - University of Michigan - Mott Children's Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Comprehensive Epilepsy Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Multicare Institute for Research and Innovation, Tacoma, Washington